CLINICAL TRIAL: NCT06151236
Title: A Phase 2, Open Label, Single Arm Clinical Trial of Neoadjuvant Nivolumab and Relatlimab in Stage I To III Resectable Merkel Cell Carcinoma
Brief Title: Neoadjuvant Nivolumab and Relatlimab in Merkel Cell Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Melanoma Institute Australia (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MIA2023/489; CA224-1064 (Other: BMS)
Record Dates: First submitted 2023-11-21; First posted 2023-11-30 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Merkel Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Merkel Cell | interventions — Nivolumab; relatlimab; Opdualag

STUDY DESIGN:
Intervention Model Description: Open label, single centre clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Neoadjuvant Treatment (Experimental): Nivolumab and relatlimab will be administered in a fixed dose combination (FDC). The FDC product contains nivolumab and relatlimab in a protein-mass ratio of 3:1 (nivolumab 240 mg and relatlimab 80 mg): in a 20 mL concentrate solution per single vial. The dose and dosing regimen for this study is nivolumab 480 mg and relatlimab 160 mg - 2 vials per infusion. This was primarily based on the observed benefit/risk profile observed in metastatic melanoma patients from Study CA224-020 pharmacokinetics (PK), pharmacodynamics, and extensive nivolumab monotherapy clinical experience. In addition, the Phase 2/3 Study CA224-047 established this dose as active in unresectable and metastatic melanoma.
  This study is open label and single arm, with all patients scheduled to receive two doses of nivolumab and relatlimab FDC prior to surgery on days 1 and 29.
  Interventions: Drug: Nivolumab 240 mg / Relatlimab 80 mg in a fixed dose combination

INTERVENTIONS:
Drug: Nivolumab 240 mg / Relatlimab 80 mg in a fixed dose combination — Dual inhibition of the distinct LAG3 and PD-1 checkpoint pathways
  Other Names: Opdualag

SUMMARY:
The goal of this clinical trial is to test neoadjuvant dual immunotherapy in Merkel cell carcinoma with the aim to improve recurrence-free survival

DETAILED DESCRIPTION:
This is a phase 2, open label, single cohort, single centre, clinical trial of neoadjuvant immunotherapy with dual inhibition of PD-1 and LAG-3 immune checkpoint pathways. The hypothesis is that neoadjuvant therapy produces a higher pathological response rate (pCR) and a longer recurrence-free survival in a cohort of treatment-naïve patients with resectable stage I (≥10 mm) to stage III Merkel cell carcinoma compared to neoadjuvant nivolumab monotherapy in Checkmate 358 (n=123, NCT02488759, historical control).

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥ 18 years
2. Written consent
3. Histologically confirmed, resectable Merkel cell carcinoma with AJCC (8th ed) clinical stage I (≥ 10 mm), IIA, or IIB or III disease
4. In-transit metastases are permitted if they are completely resectable
5. Measurable disease according to RECIST 1.1 criteria
6. Previous radiotherapy permitted if there is RECIST-measurable progression of disease since the completion of radiotherapy
7. At least one of either, archival tissue from a primary or nodal MCC lesion (if applicable) for the current diagnosis and/or a newly obtained core biopsy of a lesion which has not been previously irradiated.
8. ECOG 0-1
9. Adequate organ function on blood pathology
10. Life expectancy >12 months
11. Female patients to use effective contraception during study treatment and for 5 months after last dose.

Exclusion Criteria:

1. Clinical or radiographic evidence of distant metastases
2. Contraindication to nivolumab and / or relatlimab
3. Prior anti-PD-1, CTLA-4, PDL-1 or LAG 3 antibody exposure, or an agent directed to another stimulatory or co-inhibitory T-cell receptor for any disease or any chemotherapy or experimental local or systemic drug treatment
4. Active autoimmune disease or requirement for chronic steroid therapy other than hormone replacement therapy
5. A diagnosis of immunodeficiency or chronic steroid therapy >10 mg OD prednisone or equivalent
6. Additional malignancy active within past 3 years; patients with chronic lymphocytic leukaemia can be included in this study.
7. Uncontrolled cardiovascular disease or history of myocarditis
8. Has had an allogenic tissue/solid organ transplant
9. Troponin T (TnT) or I (TnI) >2 × institutional ULN
10. Has a history of (non-infectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis or current interstitial lung disease
11. Has an active infection requiring systemic therapy
12. Active Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or Hepatitis C virus (defined as HCV RNA [qualitative] is detected) infection.
13. Known HIV
14. Pregnant or breast feeding females
15. Concurrent medical or social conditions that may prevent the patient attending assessments or procedures per schedule

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-03-11 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2034-04 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response rate | Week 6
  Proportion of patients with a pathological complete response, as determined on the week 6 surgical specimen using the guidelines published by the International Neoadjuvant Melanoma Consortium: Complete pathological response (pCR) = 0% viable tumour cells in the surgical specimen

SECONDARY OUTCOMES:
Pathological non-complete response rate to neoadjuvant immunotherapy | Week 6
  Proportion of patients with each non-pCR response category, as determined on the week 6 surgical specimen using the guidelines published by the International Neoadjuvant Melanoma Consortium:
  * Near complete pathological response - (near pCR) - >0% - ≤10% viable tumour
  * Partial pathological response (pPR) - >10 - ≤50% viable tumour
  * Non pathological response (pNR) - >50% viable tumour
Toxicity and tolerability of neoadjuvant immunotherapy and surgical complications | Week 24
  The proportion of patients with adverse events (AE) as described in CTCAE version 5.0, from the initiation of study treatment until at least 135 days after the end of treatment. Outcome measures include the proportion of patients with:
  * An AE by CTCAE term and grade and duration
  * AEs attributable to neoadjuvant study treatment
  * Grade 3/4/5 AEs by AE term
  * A requirement to interrupt study treatment and/or delay surgery within time limit due to an AE
  * A requirement to discontinue study treatment early due to an AE
  * A requirement for oral or parenteral steroid treatment for immune-related adverse events.
  * Post-operative complications (e.g. seroma formation, wound infection or lymphoedema) and duration of events.
  * The surgeon's assessment of 'operability' from baseline and at surgery according to the INMC surgical questionnaire.
  * Clavien Dindo classification at 3, 12 and 48 weeks post surgery.
Objective response rate to neoadjuvant immunotherapy | Week 6
  The proportion of patients within each response category, as assessed using RECIST version 1.1, comparing week 6 to baseline CT and MRI.
  Objective response rate= CR and PR
Metabolic response rate to neoadjuvant immunotherapy | Week 6
  The proportion of patients within each response category, as assessed using PERCIST (standardised uptake value [SUV]) comparing week 6 to baseline PET.
  Metabolic response rate = CMR and PMR.
Recurrence-free survival | 10 years
  The proportion of patients alive and disease free from the time of surgery
Disease progression rate | Week 6
  1. The proportion of patients alive and with RECIST-defined progression of disease from the date of consent to the first radiographical evidence of local, regional or distant progression.
  2. Disease progression which leads to unresectable MCC.
Event-free survival (EFS) rate | 10 years
  The proportion of patients with EFS defined as from the time of first dose of study treatment to the earliest of:
  1. Disease progression to unresectable stage III or stage IV disease)
  2. Recurrence of MCC
  3. Treatment-related death
  4. Disease related death
Overall survival rate | 10 years
  The proportion of patients alive at years 1, 2, 5 and 10, and to actual date of death (in months), from the initiation of study treatment.
Patient reported quality of life | 1 year
  1. Changes in patient rated quality of life scores using QLQ-C30 and EQ-5D-5L from date of consent to 6 -12 weekly intervals until the end of year 1.
  2. The correlation of patient-rated quality of life scores with adverse events.
Study treatment completion rate | Week 8
  1. Proportion of patients receiving full neoadjuvant drug treatment per schedule and number of treatments missed.
  2. Proportion of patients undergoing planned surgery at week 6.
  3. Reasons for incomplete study treatment e.g. adverse event, withdrawn consent, , disease progression, patient lost to follow-up.

OTHER OUTCOMES:
Polyomavirus positivity | Week 6
  1. Proportion of patients with and without polyomavirus in tumour tissue at baseline.
  2. Correlate Merkel cell polyomavirus viral positivity (MCPyV+) in stage I-III MCC with pathological response.
Biomarkers of response, resistance, toxicity | Week 6
  * Morphological assessment H&E, including viable MCC cells, Ki67, TILs density, % fibrosis, % necrosis, compared with paired baseline measures.
  * Tumour PD-L1 expression status (+ve status = ≥1% tumour cells positive staining using Dako 28-8 PD-L1 IHC assay).
  * Characterisation of immune profile in tumour microenvironment using multiplex immunohistochemistry and Imaging mass cytometry.
  * RNA sequencing - gene expression profile including potential to perform single cell analysis on dissection specimen from tumour dissociates (single cell RNA seq).
  * Characterisation of peripheral immune profile through Cytometry by time of flight.
  * DNA sequencing to determine tumour mutational burden and key somatic mutations.
  * Response to treatment using circulating tumour DNA in peripheral blood using droplet digital PCR to quantify tumour DNA (copies/ml plasma) of known mutation in MCC tissue.
Correlation of gut microbiome on outcomes | Week 6
  1. Correlation of bacterial diversity and abundance with treatment response and incidence of treatment-related toxicities
  2. Correlation of self-reported dietary habits (including use of oral probiotics) at baseline and impact on bacterial diversity in the gut
  3. The use of antibiotics and/or steroids during neoadjuvant treatment and the impact on intestinal bacterial diversity and abundance
Correlation of outcome measures | Week 6
  Proportion of patients with concordance in pathological response, RECIST response and metabolic response (PERCIST)
Assessment of concordance between RECIST and immune-related response criteria | Week 6
  Proportion of patients with CR, PR, SD and PD as measured with both response criteria
Comparison of outcomes against CheckMate | 10 years
  Comparison of primary and secondary efficacy outcomes to those reported in the Checkmate 358 trial

CONTACTS AND LOCATIONS:
Overall Officials: Georgina V Long, Principal Investigator — Melanoma Instiute Australia
Locations (1):
- Melanoma Institute Australia, Wollstonecraft, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No